CLINICAL TRIAL: NCT02653612
Title: Intraoperative Imaging of Pulmonary Adenocarcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study has been terminated, without having enrolled any participants
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLNB-009-14F
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
Keywords: surgery; folate receptor
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): This cohort will receive the contrast agent
  Interventions: Drug: EC17 imaging contrast agent

INTERVENTIONS:
Drug: EC17 imaging contrast agent — This is an imaging agent to locate lung adenocarcinoma cancer cells during surgery

SUMMARY:
The goal is to improve surgery by preventing tumor cells from being left behind at the time of surgery. This includes finding residual tumor cells in the wound after surgery.

DETAILED DESCRIPTION:
The goal is to improve the intraoperative identification of tumor cells at positive margins and regional metastases that may be missed by a surgeon during a pulmonary resection. Improved identification of tumor cells will result in superior disease clearance and more accurate clinical staging. The investigators hypothesize that targeted fluorescent imaging during surgery will improve identification of positive margins and metastases. Since folate receptor alpha (FR ) is expressed on 55% of resectable lung cancer, the investigators will utilize a fluorescent probe that targets these tumors. As real-time imaging provides more information to the surgeon, more personalized and directed operations can be conducted. This work will allow for more preservation of normal tissue, decreased morbidity, decreased surgical time, increased surgical confidence, improved cancer detection, decreased unnecessary surgery and ultimately improved tumor free survival. This technology should transform clinical surgery from an art that depends fully on the human factor to a procedure that has precision and fail safes.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* surgical candidate
* operable
* resectable

Exclusion Criteria:

- no allergies to contrast dyes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Margin assessment | At the time of surgery
  Percentage of surgeries which detect tumor cells at the surgical margin
Lymph node assessment | 4 hours
  Number of residual tumor cells in the lymph nodes detected via intraoperative imaging of a FR-targeted fluorescent contrast agent

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Gaughan, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No